CLINICAL TRIAL: NCT04642963
Title: Stereotactic Management of Arrhythmia - Radiosurgery in Treatment of Ventricular Tachycardia
Acronym: SMART-VT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Slawomir Blamek, dr hab. n. med., Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART-VT
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Ablation; Noninvasive; Stereotactic Body Radiation Therapy; Radiosurgery; Substrate Ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Radiosurgery (Experimental): Patients with ventricular tachycardia will undergo a non-invasive cardiac radiosurgery using one fraction of 25 Gy to the arrhythmia substrate, as determined by the electrophysiological cardiac mapping.
  Interventions: Radiation: Cardiac Radiosurgery

INTERVENTIONS:
Radiation: Cardiac Radiosurgery — Non-invasive delivery of ablative radiotherapy dose to the arrhythmia substrate.
  Other Names: Stereotactic Arrhythmia Radioablation (STAR)

SUMMARY:
Prospective single-arm study investigating the safety of non-invasive cardiac radiosurgery for the treatment of ventricular tachycardia (VT).

DETAILED DESCRIPTION:
The standard of care for the treatment of Ventricular Tachycardia (VT) comprises of pharmacotherapy, ICD implantation and electrophysiology-guided catheter ablation. The treatment, however, is associated with a relatively high risk of VT recurrence. Given the limited therapeutic options and significant impact on patients quality of life, non-invasive cardiac radiosurgery has been recently gaining popularity in scientific literature as a viable alternative to salvage catheter ablations. Considering the scarcity of data from prospective trials and concern about the safety of the treatment method, this trial seeks to determine whether Stereotactic Management of Arrhythmia - Radiosurgery in Treatment of Ventricular Tachycardia (SMART-VT) meets the expected safety requirements for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with structural heart disease and implantable cardioverter defibrillator (ICD)
* Clinically significant arrhythmia with at least 3 VT episodes per month despite adequate pharmacological treatment.
* At least one episode of monomorphic VT registered in electrophysiological examination.
* Recurrent VT despite at least one prior catheter ablation and adequate pharmacotherapy OR contraindications to catheter ablation and/or pharmacotherapy (i.e., patient with medically contraindicated catheter ablation is obliged to undergo only pharmacotherapy prior to study enrollment).
* Patient must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

* Heart failure requiring inotropic treatment or mechanical assistance
* Arrhythmia due to cardiac channelopathy
* Reversible source of arrhythmia
* NYHA (New York Heart Association) stage IV hearth failure
* Hearth infarction or cardiac surgery in last 3 months
* Life expectancy <6 months
* Polymorphic VT
* Pregnancy
* Prior radiotherapy to the thoracic region (relative contraindication)
* Failure to induce VT during electrophysiological examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Acute toxicity evaluated using CTCAE v5.0 scale | 3 months
  The study aims to demonstrate the safety of the treatment method defined as 3-month observation without Grade III or higher adverse events in at least 6 out of 7 patients (1st stage), and in total in at least 9 out of 11 patients (2nd stage) with an interim safety analysis after obtaining data on primary outcome in first 7 patients.

SECONDARY OUTCOMES:
Efficacy of the treatment | 24 months
  Reduction of VT burden, ICD shocks and improvement in life quality as described by SF-36 (The Short Form Health Survey) v2 questionnaire. f eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Biochemical markers of cardiac injury | 24 months
  Intensity and dynamics of changes in cardiac-related biochemical indices after treatment, like troponin, cardiac creatine kinase (MB-CK) concentration and N-terminal prohormone of brain natriuretic peptide (NT-proBNP) to assess the early cardiac muscle damage and changes in severity of congestive heart failure.
Late toxicity and mortality | 24 months
  Assessment of late toxicity including occurrence of cardiac-related hospitalizations and death.
Anti-arrhythmic drugs uptake | 24 months
  Changes in the anti-arrhythmic medications over time after treatment.
Cardiac injury | 24 months
  Assessment of the post-treatment cardiac injury including left ventricular ejection fraction, echocardiography and morphological changes in imaging studies.
Target volume delineation | 24 months
  Correlation of electrophysiological mapping with the results of additional cardiac imaging methods (MR, PET) - only in applicable patients (optional diagnostic methods)

CONTACTS AND LOCATIONS:
Overall Officials: Sławomir Blamek, dr hab. n. med., Principal Investigator — Maria Sklodowska-Curie National Research Institute of Oncology (MSCNRIO); Wojciech Wojakowski, prof. dr hab. n. med., Principal Investigator — Upper Silesian Medical Center Professor Leszek Giec of the Medical University of Silesia in Katowice; Marcin Miszczyk, dr n. med., Study Chair — Maria Sklodowska-Curie National Research Institute of Oncology (MSCNRIO)
Locations (2):
- Poland (2):
  - Maria Sklodowska-Curie National Research Institute of Oncology (MSCNRIO), Gliwice branch, Gliwice, Silesian Voivodeship
  - Upper Silesian Medical Center Professor Leszek Giec of the Medical University of Silesia in Katowice, Katowice

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will be shared within the European STOPSTORM consortium, which is dedicated to the development of cardiac radiosurgery for the treatment of ventricular tachycardia. The intention to share anonymized data with the consortium will be clearly explained, and a written consent will be obtained from each participant.